CLINICAL TRIAL: NCT05073497
Title: The Effect of Finger Puppet on Children's Pain and Emotional Indicators Undergoing Venipuncture in Pediatric Emergency Department
Brief Title: Efficacy of Finger Puppet as a Distraction Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Zeynep Erkut, Assistant Professor, PhD, Biruni University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/51-34
Record Dates: First submitted 2021-09-18; First posted 2021-10-11 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Procedural Pain; Pain; Acute Pain
Keywords: Distraction; Finger puppet; pain management; procedural pain
MeSH Terms: conditions — Pain, Procedural; Pain; Acute Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): One minute before the procedure the children in the experimental group will start to play with finger puppets under the direction of the researcher. The researcher will continue to distract the child's attention during the procedure with finger puppets.
  Interventions: Other: Finger puppets
- Control Group (No Intervention): No intervention will perform to reduce pain in the control group.

INTERVENTIONS:
Other: Finger puppets — In the experimental group, for distraction the researcher will put finger puppets consisting of various animal figures on his finger, and will ask the child to imitate these sounds by making animal-specific sounds that he moves with his finger. The researcher will also draw the child's attention to finger puppets by using methods such as making animals talk to each other and singing before and during venipuncture.
  Arms: Experimental Group

SUMMARY:
The study will be conducted with the randomized controlled experimental method. The children who attended the pediatric emergency department will divide into two groups via randomization in the computer environment. After the randomization, children in the experimental group will play with finger puppets under the direction of the researcher during venipuncture. On the other hand, no application will perform on the children in the control group during the venipuncture. The parents will also be found next to their children in both groups during the procedure.

DETAILED DESCRIPTION:
Many different non-pharmacological methods are used to cope with negative situations such as pain, fear and anxiety caused by invasive procedures in children. One of these non-pharmacological methods is the distraction. The American Pain Society recommends the use of distraction for pain control in children. With the distraction method, the child's pain is controlled and reduced by focusing the child's attention in another direction. Video games, virtual reality glasses, listening to music, watching cartoons, blowing balloons, reading books, playing with puppet/finger puppets are used as distraction methods. The aim of this study is to determine the effect of distraction method applied with finger puppet on the child's pain level and emotional indicators in children aged 3-6 years who applied to the pediatric emergency department and underwent venous blood collection. The sample size of the study has been determined by the power analysis (G*Power 3.1.9.2), in line with the results obtained from the studies which have been conducted using a similar research method. The sample size was found to be a total of 76 children including minimum of 38 children for each group. It was estimated that case losses may occur and therefore, it was decided to conduct the study with a total of 80 children including 40 children in two groups. Information Form, Face, Legs, Activity, Cry, Consolability (FLACC) Scale, and Children's Emotional Manifestation Scale will use for data collection. Children and their parents who applied to the pediatric emergency unit will inform about the study. Information about children and their parents included in the study will ask by the researcher through face-to-face interviews and these data will record in 'Information Form' five minutes before the procedure. One minute before the procedure children in the experimental group will start to play with finger puppets under the direction of the researcher. The researcher will continue to distract the child's attention during the procedure with finger puppets. For distraction the researcher will put finger puppets consisting of various animal figures on his finger, and will ask the child to imitate these sounds by making animal-specific sounds that he moves with his finger. The researcher will also draw the child's attention to finger puppets by using methods such as making animals talk to each other and singing. Children in the control group will be given routine practices and no distraction method will be applied. Before and during venipuncture children's pain will evaluate with the FLACC Scale and their emotional status will evaluate with the Children's Emotional Manifestation Scale by the healthcare provider who performs the venipuncture procedure.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 3 and 6,
* Having body temperature at normal level (36.5-37.2oC),
* Having no disease that can cause acute or chronic pain,
* Having no auditory, mental, and neurological disability that can affect their participation,
* Having no confusion.

Exclusion Criteria:

* Being younger than 3 years old and older than 6 years old,
* Having body temperature at a higher than normal level,
* Having a disease that can cause acute or chronic pain,
* Having auditory, mental, and neurological disability that can affect their participation,
* Having confusion.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change of pain from before venipuncture to during venipuncture | Before venipuncture procedure and within 2 minutes after the venipuncture procedure
  Pain will assess by the healthcare provider who performs the venipuncture procedure with the FLACC (Face, Legs, Activity, Cry, Consolability) Scale. This scale was developed to evaluate the pain of children aged 2 months to 7 years. The child's facial expression, leg movements, activity, crying, and comfortability behaviors are evaluated in relation to pain. These five behaviors are rated with 0, 1, or 2 points. The total score of the scale ranges from 0 to 10, and a high score indicates that the child has more pain. '0' points from the scale indicate no pain, '1-3' points indicate mild pain, '4-6' points indicate moderate pain, and '7-10' points indicate severe pain.

SECONDARY OUTCOMES:
Change of emotional status from before venipuncture to during venipuncture | Before venipuncture procedure and and within 2 minutes after the venipuncture procedure
  Children's emotional status will assess by the healthcare provider who performs the venipuncture procedure with the Children's Emotional Manifestation Scale. This scale was developed to objectively evaluate children's emotional behaviors towards medical procedures. In the scale, emotional indicators are evaluated according to 5 parameters (facial expression, voice, activity, interaction, cooperation level). These five parameters are scored from 1 to 5, with the lowest '5' and the highest '25' points. A high score on the scale indicates that the child displays more negative emotional behavior during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Erkut, PhD, Principal Investigator — Maltepe University; Murat Ceylan, RN, Principal Investigator — Kartal Dr. Lütfi Kirdar City Hospital
Locations (1):
- Kartal Dr. Lütfi Kırdar City Hospital, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No